CLINICAL TRIAL: NCT05437770
Title: Effects of Low-intensity Blood-flow Restricted Exercise Compared to Standard Rehabilitation in Patients With Knee Osteoarthritis - a Randomized Controlled Trial
Brief Title: Effects of Blood-flow Restricted Exercise Compared to Standard Rehabilitation in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Southern Denmark (Other); Gigtforeningen (Other); Sygekassernes Helsefond (Other); AP Moeller Foundation (Other); Aase and Ejnar Danielsens Foundation (Other); Praksisfonen (Unknown); FAPS (Unknown)
Responsible Party: Principal Investigator, Brian Sorensen, Principal investigator and PhD student, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRS-090288
Record Dates: First submitted 2022-06-11; First posted 2022-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Blood-flow restriction; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to intervention allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR (Blood-Flow Restricted exercise) (Experimental): The BFR training intervention group will perform low load blood-flow restricted exercise. Training twice a week for 12 weeks. The group will also attend a two hours education lecture with osteoarthritis information.
  Interventions: Other: BFR (Blood-Flow Restricted exercise)
- Standard rehabilitation (Active Comparator): The standard rehabilitation group will be offered participation in the Good Life with osteoArthritis in Denmark programme (GLA:D). The programme includes supervised team group training twice a week for 8 weeks and an education lecture. The GLA:D programme will be followed by 4 weeks of team group training continuing the exercises from the GLA:D programme.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: BFR (Blood-Flow Restricted exercise) — The BFR group performs unilateral training with the knee-OA diagnosed leg first. BFR exercise is performed with a pneumatic cuff placed at the top of the thigh on the leg being trained. The cuff will be inflated to 60-80 % of the total arterial occlusion pressure (AOP). The participant will afterwards perform training of the knee extensors in a leg press exercise machine and a leg extension exercise machine with a load corresponding to 30 % of the maximal load (1RM = Repetition Maximum).
  Arms: BFR (Blood-Flow Restricted exercise)
Other: Standard rehabilitation — The GLA:D programme involves a circuit training program with four stations. Each station involves two to six exercises where the participants perform 10-15 repetitions over 2-3 sets, which depends on the participants pain- and functional level. Following the 8 weeks GLA:D programme, participants will continue 4 weeks of team group training performing similar neuromuscular lower limb exercises as for the first 8 weeks.
  Arms: Standard rehabilitation

SUMMARY:
The purpose of this study is to investigate the effect of low-intensity BFR exercise on joint pain, muscle mass, and mechanical muscle function compared to standard rehabilitering in adults with knee-OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common disease in Denmark with high socioeconomical costs. Representing the most widespread non-medical and non-operative treatment modality both internationally and in Denmark, knee-OA patients often are offered a combination of patient education, weight loss counseling and physical exercise. In Denmark the GLA:D (Good Life with osteoArthritis in Denmark) concept is a nationwide training paradigm which is a combination of education and supervised neuromuscular exercise (NEMEX). Physical exercise including conventional strength training has shown positive results on OA, however a large proportion of OA-patients are forced to refrain from this type of training to excessive joint- and muscle pain during and following the training sessions.

A more joint protecting type of training (BFR = Blood-Flow Restricted exercise), which are performed using low training load (<30% of maximum load) and with a reduced blood flow to the working muscles, has shown similar results to conventional heavy strength training. Based on these observations BFR exercise seems to represent an attractive training modality in patients with knee-OA.

The aim of the present study is to investigate the effect of low-intensity BFR exercise on joint pain, muscle mass, and mechanical muscle function compared to SR in adults with knee-OA. A second aim is to investigate if 12 weeks of training is more efficient compared to 8 weeks of training.

Patients diagnosed with knee-OA are eligible to participate. Inclusion takes place via the Institute of Sportsmedicine (ISMC), and the Department of Physical and Occupational Therapy at Bispebjerg Hospital. Patients will be called in for a preparatory examination by one of the attending physicians. At the consultation a standard clinical assessment will be performed and the participant will be examined for meeting the explicit inclusion or exclusion criteria of the study. If the participant after receiving all oral and written information wishes to participate in the study, an informed consent will be obtained. Randomization procedures will be performed. A randomized controlled trial design with two groups; 1) BFR, and 2) Standard rehabilitation. A total sample size of 95 participants are needed when assuming a 20 % dropout.

The intervention period will last 12 consecutive weeks with 2 weekly training sessions at several chosen physiotherapy clinics (standard rehabilitation) and at Bispebjerg Hospital (BFR). Participants in the standard rehabilitation group will be offered participation in the GLA:D programme supervised by GLA:D certified physiotherapists. The BFR group will be trained by instructors who are experienced in BFR exercise. Testing will take place before the intervention period, after 8 weeks of training and at the end of the intervention (12 weeks) except for the muscle biopsies which will take place before the intervention period and at the end (12 weeks). Patient-reported questionnaires will furthermore be assessed 6 months after the intervention period. Patients will be tested at Bispebjerg Hospital for a number of different outcome measures including joint- and muscle pain, functional level and mechanical muscle function (strength and muscle mass).

ELIGIBILITY:
Inclusion Criteria:

* All participants must meet the American College of Rheumatology (ACR) criteria for OA 35.
* Visible OA on X-ray pictures (Kellgren & Lawrence grade 2-3).
* Unilateral pain and functional limitation for a minimum of 3 months.
* Be able to voluntarily (i.e. unassisted) perform a 90 degrees flexion in the knee.
* Be able to perform the machine exercise (knee extension) planned for the BFR training.
* Danish-speaking.
* No longer travel planned within the intervention period.

Exclusion Criteria:

* Kellgren & Lawrence grade 4.
* Bilateral OA-symptoms.
* Prior knee- or hip alloplasty.
* Glucocorticosteroid injection in the knee within the last 6 months.
* Inflammatory arthritis.
* Known neurotic disease such as multiple sclerosis or peripheral neuropathy.
* Prior myocardial infarct or apoplexy, or chest pain during physical activity.
* Other health related or medical conditions which makes it impossible participate in the study.

Furthermore, it is an exclusion criterium in the following conditions where use of pneumatic occlusion would be considered contraindicated:

* Peripheral vascular disease
* Excessive varicose veins
* Prior history of deep venous thrombosis
* Venous insufficiency causing edema in the lower legs
* Systolic blood pressure over 160 mmHg or under 100 mmHg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - Pain subscale | Baseline (0 weeks)
  KOOS is a patient reported outcome instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Primary outcome will be an assessment of the Pain subscale as a total KOOS score has not been validated. A normalized score for the entire subscale will be calculated and reported, ranging from zero (extreme symptoms) to 100 (no symptoms).
Knee injury and Osteoarthritis Outcome Score (KOOS) - Pain subscale | 8 weeks of training.
  KOOS is a patient reported outcome instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Primary outcome will be an assessment of the Pain subscale as a total KOOS score has not been validated. A normalized score for the entire subscale will be calculated and reported, ranging from zero (extreme symptoms) to 100 (no symptoms).
Knee injury and Osteoarthritis Outcome Score (KOOS) - Pain subscale | 12 weeks of training.
  KOOS is a patient reported outcome instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Primary outcome will be an assessment of the Pain subscale as a total KOOS score has not been validated. A normalized score for the entire subscale will be calculated and reported, ranging from zero (extreme symptoms) to 100 (no symptoms).
Knee injury and Osteoarthritis Outcome Score (KOOS) - Pain subscale | 6 months after the training intervention period.
  KOOS is a patient reported outcome instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Primary outcome will be an assessment of the Pain subscale as a total KOOS score has not been validated. A normalized score for the entire subscale will be calculated and reported, ranging from zero (extreme symptoms) to 100 (no symptoms).

SECONDARY OUTCOMES:
Myofiber Cross-Sectional Area (CSA) | Baseline (0 weeks), 8 weeks and 12 weeks (the end of the intervention period)
  Quadriceps myofiber cross-sectional area will be measured using a GE Logiq E10 Logic View ultrasound to generate panoramic CSA images. Orientated in the axial-plane, the ultrasound probe is positioned perpendicularly, and a water-based gel is used to promote acoustic contact between the skin and the probe. The probe is moved manually with a slow and continuous movement from the lateral to the medial part of quadriceps along a marked line on the skin. The anatomical site for all measurements will be at 50% of the distance between the lateral condyle and greater trochanter of the femur.
Pain Pressure Threshold (PPT) | Baseline (0 weeks), 8 weeks and 12 weeks (the end of the intervention period)
  PPT is measured by a handheld pain pressure algometer at three different locations bilaterally. Most painful area in the medial joint line, tibialis anterior, and the muscle belly of extensor carpi radialis.
Maximal Voluntary Isometric Contraction (MVIC) | Baseline (0 weeks), 8 weeks and 12 weeks (the end of the intervention period)
  MVIC of the knee extensors is obtained during static knee extension in a KinCom, isokinetic dynamometer, at a knee joint angle of 70 degrees (0 degrees = full knee extension).
Rate of Force Development (RFD) | Baseline (0 weeks), 8 weeks and 12 weeks (the end of the intervention period)
  RFD of the knee extensors is obtained during static knee extension in a KinCom, isokinetic dynamometer, at a knee joint angle of 70 degrees (0 degrees = full knee extension).
4x10m Fast-Paced Walk Test (40m-FWT) | At baseline (0 weeks), 8 weeks, 12 weeks (the end of the intervention period)
  The 40m-FWT is a test of walking speed over short distances and changing direction during walking. It measures the total time it takes to walk 4 * 10 m excluding turns (m/s).
30-second Chair Stand Test (30-s CST) | At baseline (0 weeks), 8 weeks, 12 weeks (the end of the intervention period).
  The 30-s CST is used for testing leg strength and endurance. The 30-s CST will be assessed using a chair (seat height: 43-44 cm) with armrests. The 30-s CST measures the number of sit-to-stand repetitions completed within 30-s.
Stair Climb Test (SCT) | At baseline (0 weeks), 8 weeks, 12 weeks (the end of the intervention period).
  The SCT involves ascending and descending 10 stairs measuring 18 cm rise / 92 cm width. Each participant is asked to ascend/descend the stairs at their ''natural'' pace (without resting). One trial to ascend and descend is timed and recorded electronically.
Myocellular component (Stem cells) assessed using muscle biopsies | Baseline (0 weeks) and 12 weeks (the end of the intervention period)
  Muscle biopsies will be obtained for determination of important myocellular components (number of muscular stem cells). It will be assessed by obtaining needle biopsies (100-150 mg). The biopsies will be obtained unilaterally from the middle portion of the vastus lateralis muscle using the percutaneous needle biopsy technique of Bergström.
Myocellular component (Fiber area) assessed using muscle biopsies | Baseline (0 weeks) and 12 weeks (the end of the intervention period)
  Muscle biopsies will be obtained for determination of important myocellular components (fiber area in diameter: μm2). It will be assessed by obtaining needle biopsies (100-150 mg). The biopsies will be obtained unilaterally from the middle portion of the vastus lateralis muscle using the percutaneous needle biopsy technique of Bergström.
Myocellular component (Myonuclei) assessed using muscle biopsies | Baseline (0 weeks) and 12 weeks (the end of the intervention period)
  Muscle biopsies will be obtained for determination of important myocellular components (number of myonuclei). It will be assessed by obtaining needle biopsies (100-150 mg). The biopsies will be obtained unilaterally from the middle portion of the vastus lateralis muscle using the percutaneous needle biopsy technique of Bergström.
Maximal lower limb muscle power | Baseline (0 weeks), 8 weeks and 12 weeks (the end of the intervention period)
  Explosive lower limb muscle power will be assessed during a single-legged extensor power-rig. Subjects will be seated in the power-rig chair and pushes away the footplate connected to a flywheel as hard and fast as possible.
Knee injury and Osteoarthritis Outcome Score (KOOS) | At baseline (0 weeks), 8 weeks, 12 weeks (the end of the intervention period) and 6 months after the intervention period.
  KOOS is a patient reported outcome instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). A normalized score for the total KOOS score will be calculated and reported, ranging from zero (extreme symptoms) to 100 (no symptoms).
Oxford Knee Score | At baseline (0 weeks), 8 weeks, 12 weeks (the end of the intervention period) and 6 months after the intervention period.
  The Oxford Knee Score is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks. Each question is scored from 0-4 where four is the best outcome and total scores range from 0 (poorest function) to 48 (maximal function).

CONTACTS AND LOCATIONS:
Overall Officials: Finn E Johannsen, MD, Principal Investigator — Institute of Sports Medicine
Locations (1):
- Department of Physical and Occupational Therapy / Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverwood V, Blagojevic-Bucknall M, Jinks C, Jordan JL, Protheroe J, Jordan KP. Current evidence on risk factors for knee osteoarthritis in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Apr;23(4):507-15. doi: 10.1016/j.joca.2014.11.019. Epub 2014 Nov 29. PMID 25447976
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Background] Dantas LO, Salvini TF, McAlindon TE. Knee osteoarthritis: key treatments and implications for physical therapy. Braz J Phys Ther. 2021 Mar-Apr;25(2):135-146. doi: 10.1016/j.bjpt.2020.08.004. Epub 2020 Sep 8. PMID 33262080
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Holm PM, Schroder HM, Wernbom M, Skou ST. Low-dose strength training in addition to neuromuscular exercise and education in patients with knee osteoarthritis in secondary care - a randomized controlled trial. Osteoarthritis Cartilage. 2020 Jun;28(6):744-754. doi: 10.1016/j.joca.2020.02.839. Epub 2020 Mar 13. PMID 32179197
- [Background] Skou ST, Rasmussen S, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Roos EM. The efficacy of 12 weeks non-surgical treatment for patients not eligible for total knee replacement: a randomized controlled trial with 1-year follow-up. Osteoarthritis Cartilage. 2015 Sep;23(9):1465-75. doi: 10.1016/j.joca.2015.04.021. Epub 2015 Apr 30. PMID 25937024
- [Background] Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. J Rheumatol. 2014 Jul;41(7):1385-94. doi: 10.3899/jrheum.130642. Epub 2014 Jun 15. PMID 24931956
- [Background] Roos EM, Gronne DT, Skou ST, Zywiel MG, McGlasson R, Barton CJ, Kemp JL, Crossley KM, Davis AM. Immediate outcomes following the GLA:D(R) program in Denmark, Canada and Australia. A longitudinal analysis including 28,370 patients with symptomatic knee or hip osteoarthritis. Osteoarthritis Cartilage. 2021 Apr;29(4):502-506. doi: 10.1016/j.joca.2020.12.024. Epub 2021 Feb 6. PMID 33561542
- [Background] Skou ST, Odgaard A, Rasmussen JO, Roos EM. Group education and exercise is feasible in knee and hip osteoarthritis. Dan Med J. 2012 Dec;59(12):A4554. PMID 23290290
- [Background] Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. BMC Musculoskelet Disord. 2017 Feb 7;18(1):72. doi: 10.1186/s12891-017-1439-y. PMID 28173795
- [Background] Bennell KL, Hunt MA, Wrigley TV, Lim BW, Hinman RS. Role of muscle in the genesis and management of knee osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):731-54. doi: 10.1016/j.rdc.2008.05.005. PMID 18687280
- [Background] Skoffer B, Dalgas U, Mechlenburg I, Soballe K, Maribo T. Functional performance is associated with both knee extensor and flexor muscle strength in patients scheduled for total knee arthroplasty: A cross-sectional study. J Rehabil Med. 2015 May;47(5):454-9. doi: 10.2340/16501977-1940. PMID 25678417
- [Background] Bryk FF, Dos Reis AC, Fingerhut D, Araujo T, Schutzer M, Cury Rde P, Duarte A Jr, Fukuda TY. Exercises with partial vascular occlusion in patients with knee osteoarthritis: a randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1580-6. doi: 10.1007/s00167-016-4064-7. Epub 2016 Mar 12. PMID 26971109
- [Background] Ferraz RB, Gualano B, Rodrigues R, Kurimori CO, Fuller R, Lima FR, DE Sa-Pinto AL, Roschel H. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. Med Sci Sports Exerc. 2018 May;50(5):897-905. doi: 10.1249/MSS.0000000000001530. PMID 29266093
- [Background] Manimmanakorn A, Hamlin MJ, Ross JJ, Taylor R, Manimmanakorn N. Effects of low-load resistance training combined with blood flow restriction or hypoxia on muscle function and performance in netball athletes. J Sci Med Sport. 2013 Jul;16(4):337-42. doi: 10.1016/j.jsams.2012.08.009. Epub 2012 Sep 19. PMID 22999393
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Blood flow restricted exercise for athletes: A review of available evidence. J Sci Med Sport. 2016 May;19(5):360-7. doi: 10.1016/j.jsams.2015.04.014. Epub 2015 May 9. PMID 26118847
- [Background] Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. Br J Sports Med. 2017 Dec;51(23):1688-1694. doi: 10.1136/bjsports-2016-096329. Epub 2017 May 12. PMID 28500081
- [Background] Gronfeldt BM, Lindberg Nielsen J, Mieritz RM, Lund H, Aagaard P. Effect of blood-flow restricted vs heavy-load strength training on muscle strength: Systematic review and meta-analysis. Scand J Med Sci Sports. 2020 May;30(5):837-848. doi: 10.1111/sms.13632. Epub 2020 Feb 21. PMID 32031709
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. J Appl Physiol (1985). 2020 Apr 1;128(4):914-924. doi: 10.1152/japplphysiol.00768.2019. Epub 2020 Feb 27. PMID 32105522
- [Background] Lixandrao ME, Ugrinowitsch C, Berton R, Vechin FC, Conceicao MS, Damas F, Libardi CA, Roschel H. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. Sports Med. 2018 Feb;48(2):361-378. doi: 10.1007/s40279-017-0795-y. PMID 29043659
- [Background] Takada S, Okita K, Suga T, Omokawa M, Kadoguchi T, Sato T, Takahashi M, Yokota T, Hirabayashi K, Morita N, Horiuchi M, Kinugawa S, Tsutsui H. Low-intensity exercise can increase muscle mass and strength proportionally to enhanced metabolic stress under ischemic conditions. J Appl Physiol (1985). 2012 Jul;113(2):199-205. doi: 10.1152/japplphysiol.00149.2012. Epub 2012 May 24. PMID 22628373
- [Background] Yasuda T, Fukumura K, Fukuda T, Uchida Y, Iida H, Meguro M, Sato Y, Yamasoba T, Nakajima T. Muscle size and arterial stiffness after blood flow-restricted low-intensity resistance training in older adults. Scand J Med Sci Sports. 2014 Oct;24(5):799-806. doi: 10.1111/sms.12087. Epub 2013 Jun 3. PMID 23730848
- [Background] Dos Santos LP, Santo RCDE, Ramis TR, Portes JKS, Chakr RMDS, Xavier RM. The effects of resistance training with blood flow restriction on muscle strength, muscle hypertrophy and functionality in patients with osteoarthritis and rheumatoid arthritis: A systematic review with meta-analysis. PLoS One. 2021 Nov 10;16(11):e0259574. doi: 10.1371/journal.pone.0259574. eCollection 2021. PMID 34758045
- [Background] Rodrigues R, Ferraz RB, Kurimori CO, Guedes LK, Lima FR, de Sa-Pinto AL, Gualano B, Roschel H. Low-Load Resistance Training With Blood-Flow Restriction in Relation to Muscle Function, Mass, and Functionality in Women With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2020 Jun;72(6):787-797. doi: 10.1002/acr.23911. Epub 2020 May 14. PMID 31033228
- [Background] Centner C, Wiegel P, Gollhofer A, Konig D. Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. Sports Med. 2019 Jan;49(1):95-108. doi: 10.1007/s40279-018-0994-1. PMID 30306467
- [Background] Nielsen JL, Aagaard P, Bech RD, Nygaard T, Hvid LG, Wernbom M, Suetta C, Frandsen U. Proliferation of myogenic stem cells in human skeletal muscle in response to low-load resistance training with blood flow restriction. J Physiol. 2012 Sep 1;590(17):4351-61. doi: 10.1113/jphysiol.2012.237008. Epub 2012 Jul 16. PMID 22802591
- [Background] Ramos-Campo DJ, Scott BR, Alcaraz PE, Rubio-Arias JA. The efficacy of resistance training in hypoxia to enhance strength and muscle growth: A systematic review and meta-analysis. Eur J Sport Sci. 2018 Feb;18(1):92-103. doi: 10.1080/17461391.2017.1388850. Epub 2017 Oct 18. PMID 29045191
- [Background] Jakobsgaard JE, Christiansen M, Sieljacks P, Wang J, Groennebaek T, de Paoli F, Vissing K. Impact of blood flow-restricted bodyweight exercise on skeletal muscle adaptations. Clin Physiol Funct Imaging. 2018 Feb 15. doi: 10.1111/cpf.12509. Online ahead of print. PMID 29446524
- [Background] Kubo K, Komuro T, Ishiguro N, Tsunoda N, Sato Y, Ishii N, Kanehisa H, Fukunaga T. Effects of low-load resistance training with vascular occlusion on the mechanical properties of muscle and tendon. J Appl Biomech. 2006 May;22(2):112-9. doi: 10.1123/jab.22.2.112. PMID 16871002
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Clarkson MJ, May AK, Warmington SA. Is there rationale for the cuff pressures prescribed for blood flow restriction exercise? A systematic review. Scand J Med Sci Sports. 2020 Aug;30(8):1318-1336. doi: 10.1111/sms.13676. Epub 2020 Apr 27. PMID 32279391
- [Background] Patterson SD, Hughes L, Head P, Warmington S, Brandner C. Blood flow restriction training: a novel approach to augment clinical rehabilitation: how to do it. Br J Sports Med. 2017 Dec;51(23):1648-1649. doi: 10.1136/bjsports-2017-097738. Epub 2017 Jun 22. No abstract available. PMID 28642225
- [Background] Næss, T.C. (2021). Determining the optimal blood flow restriction protocol for maximising muscle hypertrophy and strength, pressure and cuff width: A mini-review. Journal of Human Sport and Exercise, 16(4), 752-759
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Vanwye WR, Weatherholt AM, Mikesky AE. Blood Flow Restriction Training: Implementation into Clinical Practice. Int J Exerc Sci. 2017 Sep 1;10(5):649-654. doi: 10.70252/LYGQ7085. eCollection 2017. PMID 28966705
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Sturnieks DL, Arnold R, Lord SR. Validity and reliability of the Swaymeter device for measuring postural sway. BMC Geriatr. 2011 Oct 20;11:63. doi: 10.1186/1471-2318-11-63. PMID 22011335
- [Background] Suetta C, Magnusson SP, Rosted A, Aagaard P, Jakobsen AK, Larsen LH, Duus B, Kjaer M. Resistance training in the early postoperative phase reduces hospitalization and leads to muscle hypertrophy in elderly hip surgery patients--a controlled, randomized study. J Am Geriatr Soc. 2004 Dec;52(12):2016-22. doi: 10.1111/j.1532-5415.2004.52557.x. PMID 15571536
- [Background] Suetta C, Aagaard P, Rosted A, Jakobsen AK, Duus B, Kjaer M, Magnusson SP. Training-induced changes in muscle CSA, muscle strength, EMG, and rate of force development in elderly subjects after long-term unilateral disuse. J Appl Physiol (1985). 2004 Nov;97(5):1954-61. doi: 10.1152/japplphysiol.01307.2003. Epub 2004 Jul 9. PMID 15247162
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. J Appl Physiol (1985). 2002 Oct;93(4):1318-26. doi: 10.1152/japplphysiol.00283.2002. PMID 12235031
- [Background] Caserotti P, Aagaard P, Larsen JB, Puggaard L. Explosive heavy-resistance training in old and very old adults: changes in rapid muscle force, strength and power. Scand J Med Sci Sports. 2008 Dec;18(6):773-82. doi: 10.1111/j.1600-0838.2007.00732.x. Epub 2008 Jan 30. PMID 18248533
- [Background] Mertz KH, Reitelseder S, Jensen M, Lindberg J, Hjulmand M, Schucany A, Binder Andersen S, Bechshoeft RL, Jakobsen MD, Bieler T, Beyer N, Lindberg Nielsen J, Aagaard P, Holm L. Influence of between-limb asymmetry in muscle mass, strength, and power on functional capacity in healthy older adults. Scand J Med Sci Sports. 2019 Dec;29(12):1901-1908. doi: 10.1111/sms.13524. Epub 2019 Aug 16. PMID 31353627
- [Background] Nielsen JL, Frandsen U, Jensen KY, Prokhorova TA, Dalgaard LB, Bech RD, Nygaard T, Suetta C, Aagaard P. Skeletal Muscle Microvascular Changes in Response to Short-Term Blood Flow Restricted Training-Exercise-Induced Adaptations and Signs of Perivascular Stress. Front Physiol. 2020 Jun 12;11:556. doi: 10.3389/fphys.2020.00556. eCollection 2020. PMID 32595516
- [Background] Ashkavand Z, Malekinejad H, Vishwanath BS. The pathophysiology of osteoarthritis. Journal of Pharmacy Research. 2013/01/01/ 2013;7(1):132-138.
- [Background] Jensen H, Davidsen M, Ekholm O, Christensen A. Danskernes Sundhed - Den Nationale Sundhedsprofil 2021. Sundhedsstyrelsen. 2022
- [Background] Johnsen N, Kock M, Davidsen M, Juel K. De samfundsmæssige omkostninger ved artrose. Statens Institut for Folkesundhed. 2014
- [Background] Sundhedsstyrelsen. Knæartrose - Nationale kliniske retningslinjer og faglige visitationsretningslinjer. 2012
- [Background] Oiestad BE, Juhl CB, Eitzen I, Thorlund JB. Knee extensor muscle weakness is a risk factor for development of knee osteoarthritis. A systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Feb;23(2):171-7. doi: 10.1016/j.joca.2014.10.008. Epub 2014 Nov 1. PMID 25450853
- [Background] Bandak E, Christensen R, Overgaard A, Kristensen LE, Ellegaard K, Guldberg-Moller J, Bartholdy C, Hunter DJ, Altman R, Bliddal H, Henriksen M. Exercise and education versus saline injections for knee osteoarthritis: a randomised controlled equivalence trial. Ann Rheum Dis. 2022 Apr;81(4):537-543. doi: 10.1136/annrheumdis-2021-221129. Epub 2021 Nov 29. PMID 34844929
- [Background] Davis AM, Kennedy D, Wong R, Robarts S, Skou ST, McGlasson R, Li LC, Roos E. Cross-cultural adaptation and implementation of Good Life with osteoarthritis in Denmark (GLA:D): group education and exercise for hip and knee osteoarthritis is feasible in Canada. Osteoarthritis Cartilage. 2018 Feb;26(2):211-219. doi: 10.1016/j.joca.2017.11.005. Epub 2017 Nov 13. PMID 29146385
- [Background] Holm PM, Petersen KK, Wernbom M, Schroder HM, Arendt-Nielsen L, Skou ST. Strength training in addition to neuromuscular exercise and education in individuals with knee osteoarthritis-the effects on pain and sensitization. Eur J Pain. 2021 Oct;25(9):1898-1911. doi: 10.1002/ejp.1796. Epub 2021 Jun 8. PMID 33991370
- [Background] Skou ST, Bricca A, Roos EM. The impact of physical activity level on the short- and long-term pain relief from supervised exercise therapy and education: a study of 12,796 Danish patients with knee osteoarthritis. Osteoarthritis Cartilage. 2018 Nov;26(11):1474-1478. doi: 10.1016/j.joca.2018.07.010. Epub 2018 Aug 2. PMID 30076884
- [Background] Rodriguez-Lopez C, Beckwee D, Luyten FP, Van Assche D, Van Roie E. Reduced knee extensor torque production at low to moderate velocities in postmenopausal women with knee osteoarthritis. Scand J Med Sci Sports. 2021 Nov;31(11):2144-2155. doi: 10.1111/sms.14035. Epub 2021 Aug 25. PMID 34409660
- [Background] Culvenor AG, Ruhdorfer A, Juhl C, Eckstein F, Oiestad BE. Knee Extensor Strength and Risk of Structural, Symptomatic, and Functional Decline in Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Arthritis Care Res (Hoboken). 2017 May;69(5):649-658. doi: 10.1002/acr.23005. PMID 27563843
- [Background] Jan MH, Lin JJ, Liau JJ, Lin YF, Lin DH. Investigation of clinical effects of high- and low-resistance training for patients with knee osteoarthritis: a randomized controlled trial. Phys Ther. 2008 Apr;88(4):427-36. doi: 10.2522/ptj.20060300. Epub 2008 Jan 24. PMID 18218827

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT05437770/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT05437770/SAP_001.pdf